CLINICAL TRIAL: NCT04154644
Title: Performance, Safety, and Efficacy of a New Cryotherapy Device for Cervical Dysplasia
Brief Title: Performance, Safety, and Efficacy of a New Cryotherapy Device for Cervical Dysplasia [Part II]
Acronym: CryoPop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Jawaharlal Nehru Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1UH3CA189923-01
Record Dates: First submitted 2019-10-29; First posted 2019-11-06 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Cervical Dysplasia
Keywords: Cryotherapy
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cervical Cytology (Experimental): 100 women with abnormal cervical cytology will receive cryotherapy with the experimental CryoPop device
  Interventions: Device: CryoPop

INTERVENTIONS:
Device: CryoPop — The new CryoPop device will be tested on women with abnormal cytology. Benchmark testing occurred in the previous study and CryoPop was found to be non-inferior to standard cryotherapy device (MedGyn) in woman with normal cytology.

SUMMARY:
Globally, cervical cancer is the second most common cancer for women and kills approximately 250,000 women every year, with the annual number of deaths expected to increase to 410,000 by 2030. The majority (88%) of these deaths occur in low- and middle-income countries (LMICs) where screening and prevention services are limited. Prevention of cervical cancer by identification and treatment of cervical cancer precursors is key, since treatment resources for invasive disease are scarce. A cervical cancer screening program cannot be effective unless it is linked with a proven intervention to prevent the development of cervical cancer. The World Health Organization (WHO) recently released the WHO guidelines for screening and treatment of precancerous lesions for cervical cancer prevention, which recommends a screen-and-treat approach for cervical cancer prevention, with cryotherapy being the first choice of treatment for women who have a positive screen. However, these programs are still slow to be implemented in part due to the current high cost and low efficiency of cryotherapy equipment that is often prone to breaking. Jhpiego, an affiliate of Johns Hopkins University (JHU), has developed a new cryotherapy device, CryoPop, that is one tenth the cost of current equipment while also ten times more efficient. Once proven safe, feasible and effective, CryoPop could save tens of thousands of lives in low- and middle-income countries each year by preventing cervical cancer.

DETAILED DESCRIPTION:
The World Health Organization (WHO) Guidelines for screening and treatment of precancerous lesions for cervical cancer prevention recommends a screen- and-treat approach for cervical cancer prevention, with cryotherapy being the first choice of treatment for women who have a positive screen. Cryotherapy using nitrous oxide (N2O) or carbon dioxide (CO2) to induce cryonecrosis of dysplastic tissues followed by regeneration of normal cervical epithelium is the most common intervention used in LMICs because it is simple and safe enough for competently-trained mid-level providers such as nurses and midwives to operate, and can be performed without anesthesia or electricity. Adverse effects after cryotherapy are relatively uncommon and generally minor, reported in 1-2% of women. A recent meta-analysis of 77 studies (with moderate to high quality evidence) regarding the effectiveness of cryotherapy found cure rates of 92% and 85%, respectively, in CIN 2 and CIN 3. Cure was defined as normal cytology or disease-free state (generally with colposcopy +/- biopsy) at the follow-up visit, implying absence of persistent disease or recurrent lesions after treatment and length of follow-up varied from 3 months to 10 years. A more recent systematic review and meta-analyses of benefits and harms of cryotherapy, as well as Loop Electrosurgical Excision Procedure (LEEP) and cervical conization (167 studies) found a residual/ recurrence rate of cervical dysplasia (CIN 2-3) of 5% at 12 months' follow-up. Major and minor adverse events occurred in less than 1% of women and were fewer with cryotherapy than with the other approaches. Limited data suggests that preterm delivery in subsequent pregnancy may be increased (<2%) with cryotherapy or LEEP.

Cost, reliability, durability, portability and reparability are all factors that prohibit the scale-up necessary for current cryotherapy methods to match the volume of population-based screening needed to achieve a marked decrease in cervical cancer morbidity and mortality. Each cryotherapy unit costs approximately $2,000-$7500, resulting in approximately 80% or more of the treatment cost of cryotherapy being directly attributed to equipment cost. The design involves many custom parts available only through the manufacturers, which are all based in the US or Europe. This prohibits local repairs and limits the life of the product to only one or two years (or even less when spare parts are not available). Additionally, the current technology requires huge amount of N20 or CO2 requiring large gas cylinders which are heavy and costly-the cost to refill a CO2 tank can be up to $200.

The subject of this proposal, CryoPop, is a new technology specifically designed for LMIC settings and more appropriate to support see-and-treat efforts because of its low cost, portability, reparability and durability. The CryoPop device is currently expected to cost one half of the price of current devices while also using one tenth of the CO2 supply, thereby substantially reducing the recurring cost of refilling a smaller and more portable gas supply with far greater efficiency in the use of CO2. Moreover, this device is designed to have minimal moving components which at the same time are inexpensive to replace and easy to repair in- situ by the providers themselves. Finally, the CryoPop is not tethered to the gas canister during the procedure, adding more safety to the treatment procedure by not having to be concerned over tank or gas line placement.The goal is to have a device for the frontline where screening is happening and provide the unique opportunity of minimizing if not preventing loss to follow-up of screen-positive women.

This will accelerate access to cervical cancer prevention and treatment services by enabling implementation of single-visit approach (SVA) to rural, underdeveloped regions, most of which have never had cervical cancer prevention (CECAP) programs.

This clinical trial is Part 2 of a 2-part research study. Part 1 of this research study is registered under:

1UH2CA189923-01 Performance, Safety, and Efficacy of a New Cryotherapy Device for Cervical Dysplasia NCT02367625

ELIGIBILITY:
Inclusion Criteria:

1. Must be 30-49 years old
2. High-grade squamous intraepithelial lesion of the cervix (CIN 2/3), confirmed on histology
3. Eligible for cryotherapy based on size of lesion (occupies <75% of cervix) and fully visible on colposcopy or visual inspection with acetic acid (VIA)
4. Willing and able to provide consent.

Exclusion Criteria:

1. Menopausal
2. History of hysterectomy
3. Known HIV+ or active cervical infections
4. Lesion occupies >75% of cervix and/or extends into the endo cervical canal
5. Pregnancy

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of CryoPop: negative Pap smear and negative biopsy (if performed) on each study participant. | 6 months
  The proportion of pap smears and colposcopy/biopsies that are negative (have no dysplasia or cancer) as confirmed by Pap smear and/or biopsy read by 2 or 3 pathologists. If there is discordance between the Pap and biopsy readings, the reading with the greater abnormality will have priority as an endpoint.

SECONDARY OUTCOMES:
Safety of CryoPop: Incidences of adverse events documented throughout the study. | 6 months
  Percent of adverse events (AE) and serious adverse events (SAE) will be reported for the study sample. These values will be compared to the safety profile reported for another standard commercially available cryotherapy device.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Anderson, MD, Principal Investigator — janders@jhmi.edu
Locations (1):
- JN Medical College, Belagavi, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
Data and research materials will be made available for public access upon the completion of the data collection. This data will be shared through the JHU Data Archive, which uses an established repository platform (Dataverse) and is supported by preservation practices, with administrative help for preparing deposits provided by Johns Hopkins Data Services. Deposited data is given standard data citations and persistent identifiers (DOIs) and will be archived for a minimum of 5 years, with the possibility of renewal.

REFERENCES:
- [Background] Thomas G. Are we making progress in curing advanced cervical cancer? J Clin Oncol. 2011 May 1;29(13):1654-6. doi: 10.1200/JCO.2010.34.1966. Epub 2011 Mar 28. No abstract available. PMID 21444860
- [Background] Sawaya GF, Grimes DA. New technologies in cervical cytology screening: a word of caution. Obstet Gynecol. 1999 Aug;94(2):307-10. doi: 10.1016/s0029-7844(99)00289-6. PMID 10432148
- [Background] van der Graaf Y, Klinkhamer PJ, Vooijs GP. Effect of population screening for cancer of the uterine cervix in Nijmegen, The Netherlands. Prev Med. 1986 Nov;15(6):582-90. doi: 10.1016/0091-7435(86)90063-0. PMID 3797390
- [Background] Sankaranarayanan R, Rajkumar R, Esmy PO, Fayette JM, Shanthakumary S, Frappart L, Thara S, Cherian J. Effectiveness, safety and acceptability of 'see and treat' with cryotherapy by nurses in a cervical screening study in India. Br J Cancer. 2007 Mar 12;96(5):738-43. doi: 10.1038/sj.bjc.6603633. Epub 2007 Feb 20. PMID 17311015
- [Background] Nene BM, Hiremath PS, Kane S, Fayette JM, Shastri SS, Sankaranarayanan R. Effectiveness, safety, and acceptability of cryotherapy by midwives for cervical intraepithelial neoplasia in Maharashtra, India. Int J Gynaecol Obstet. 2008 Dec;103(3):232-6. doi: 10.1016/j.ijgo.2008.07.016. Epub 2008 Sep 24. PMID 18817909
- [Background] Sauvaget C, Muwonge R, Sankaranarayanan R. Meta-analysis of the effectiveness of cryotherapy in the treatment of cervical intraepithelial neoplasia. Int J Gynaecol Obstet. 2013 Mar;120(3):218-23. doi: 10.1016/j.ijgo.2012.10.014. Epub 2012 Dec 22. PMID 23265830
- [Background] Santesso N, Mustafa RA, Wiercioch W, Kehar R, Gandhi S, Chen Y, Cheung A, Hopkins J, Khatib R, Ma B, Mustafa AA, Lloyd N, Wu D, Broutet N, Schunemann HJ. Systematic reviews and meta-analyses of benefits and harms of cryotherapy, LEEP, and cold knife conization to treat cervical intraepithelial neoplasia. Int J Gynaecol Obstet. 2016 Mar;132(3):266-71. doi: 10.1016/j.ijgo.2015.07.026. Epub 2015 Nov 28. PMID 26643302
- [Background] Quentin W, Adu-Sarkodie Y, Terris-Prestholt F, Legood R, Opoku BK, Mayaud P. Costs of cervical cancer screening and treatment using visual inspection with acetic acid (VIA) and cryotherapy in Ghana: the importance of scale. Trop Med Int Health. 2011 Mar;16(3):379-89. doi: 10.1111/j.1365-3156.2010.02722.x. Epub 2011 Jan 9. PMID 21214692
- [Derived] Yogeshkumar S, Anderson J, Lu E, Kenyi E, Mensa M, Thaler K, Antartani R, Donimath K, Patil B, Chikaraddi S, Bidri S, Biradar A, Gudadinni MR, Lokare L, Yenokyan G, Bellad MB, Goudar SS, Derman R, Revankar A, Patil H, Wani R, Kangle R, Chavan RY, Nagmoti MB, Kabadi YM, Reddy P, Vernekar S, Hipparagi S, Patil V, Dalal A. Safety and efficacy of the new CryoPop(R) cryotherapy device for cervical dysplasia in low- and middle-income countries: study protocol for a multicenter open-label non-inferiority clinical trial with historical controls. Trials. 2021 Dec 13;22(1):915. doi: 10.1186/s13063-021-05802-8. PMID 34903244
- See also: WHO guidelines for screening and treatment of precancerous lesions for cervical cancer prevention — https://apps.who.int/iris/bitstream/handle/10665/94830/9789241548694_eng.pdf;sequence=1